CLINICAL TRIAL: NCT00931112
Title: Effects of Individualized Exercise Training on Arterial Function, Walking Ability and Quality of Life in Patients With Peripheral Arterial Disease Post Surgery
Brief Title: Effects of Individualized Exercise Training in Patients With Peripheral Arterial Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Ying-Tai Wu, National Taiwan University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 9561709137
Record Dates: First submitted 2009-07-01; First posted 2009-07-02 (Estimated); Last update posted 2009-07-22 (Estimated); Status verified 2009-07

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral Arterial Disease; Walking ability; Quality of life; Exercise training
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- exercise (Other)
  Interventions: Other: individualized exercise training

INTERVENTIONS:
Other: individualized exercise training — Lower extremities resistance exercise and bicycle training
  Other Names: exercise

SUMMARY:
The study is designed to investigate individualized exercise training effects on arterial function, walking ability and quality of life in subjects with peripheral arterial disease post surgery.

ELIGIBILITY:
Inclusion Criteria:

* Peripheral arterial disease post surgery > 1 month
* No discharge of surgical incision
* Intermittent claudication post invasive treatment

Exclusion Criteria:

* Necrosis
* Above/below knee amputee
* Other conditions might affect peripheral vascular elasticity

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2006-11; Primary Completion 2007-05 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
arterial function, walking ability and quality of life | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan